CLINICAL TRIAL: NCT05654883
Title: New York City Observational Study of Mpox Immunity: NYC OSMI
Brief Title: New York City Observational Study of Mpox Immunity
Acronym: NYC OSMI
Status: Enrolling by invitation | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 22-01338
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Monkeypox; Mpox; HIV
Keywords: Vaccine; Immunity; Intradermal
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (11):
- HIV-negative, SQ-SQ, short interval: HIV-negative patients who received two subcutaneous mpox vaccinations with an interval of <7 weeks between primer and booster doses.
- HIV-positive, SQ-SQ, short interval: HIV-positive patients who received two subcutaneous mpox vaccinations with an interval of <7 weeks between primer and booster doses.
- HIV-negative, ID-ID, short interval: HIV-negative patients who received two intradermal mpox vaccinations with an interval of <7 weeks between primer and booster doses.
- HIV-positive, ID-ID, short interval: HIV-positive patients who received two intradermal mpox vaccinations with an interval of <7 weeks between primer and booster doses.
- HIV-negative, SQ-SQ, SQ-ID, ID-SQ or ID-ID, long interval: HIV-negative patients who received either:
  1. subcutaneous primer and booster mpox vaccinations, OR
  2. intradermal primer and booster mpox vaccinations, OR
  3. subcutaneous primer followed by intradermal booster mpox vaccination OR
  4. intradermal primer followed by subcutaneous booster mpox vaccination
  with the booster dose being taken after an interval of ≥7 weeks.
- HIV-positive, SQ-SQ, SQ-ID, ID-SQ or ID-ID, long interval: HIV-positive patients who received either:
  1. subcutaneous primer and booster mpox vaccinations, OR
  2. intradermal primer and booster mpox vaccinations, OR
  3. subcutaneous primer followed by intradermal booster mpox vaccination OR
  4. intradermal primer followed by subcutaneous booster mpox vaccination
  with the booster dose being taken after an interval of ≥7 weeks.
- SQ-ID or ID-SQ, short interval: 1. subcutaneous primer and intradermal booster mpox vaccinations, OR
  2. intradermal primer and subcutaneous booster mpox vaccinations
  with the booster dose being taken after an interval of <7 weeks.
- 1st Dose Only: Participants who receive a 1st dose of the mpox vaccination but elect not to take 2nd dose.
- Convalescent, No Vaccination: Participants who are convalescent from mpox infection who do not receive mpox vaccination.
- Convalescent, Vaccination Post-Infection: Participants who are convalescent from mpox infection who receive mpox vaccination after infection.
- BT after Vaccinations: Participants who experienced breakthrough (BT) mpox infections following mpox vaccination.

SUMMARY:
The goal of this study is to assess the immune response, tolerance, and safety of the low-dose intradermal (forearm) mpox vaccine in people who are HIV+ compared to people who are HIV-, and compared to the standard-dose subcutaneous (upper arm) vaccine. The resulting data will fill knowledge gaps, inform public health practices, and address community concerns about the absence of data for low-dose intradermal mpox vaccinations in people living with HIV.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to understand and sign the Informed Consent Form (ICF)
2. ≥18 years of age

   a. Including breastfeeding and pregnant people
3. Must have one or the other of criteria a and b, or can have both:

   1. Planning receipt of (in the next 30 days) or have received the mpox vaccine, and/or
   2. people with recent mpox infection who are out of isolation (≥30 days after symptom onset)
4. Willingness and ability to participate in all study procedures

Exclusion Criteria:

1. Known clinically significant anemia (i.e., Hb < 10 g/dL)
2. Contraindication to phlebotomy based on investigator judgement; e.g., anti-coagulation therapy with history of phlebotomy complications, or clinically significant thrombocytopenia
3. Any condition that, in the opinion of the Investigator, would make study participation unsafe for the individual or would interfere with the objectives of the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The NYC OSMI observational cohort will be drawn from NYC communities within the broad Vaccine Center catchment area.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Geometric Mean Titer (GMT) of Serum Neutralization of Mpox Virus approximately 14 Days After Second Vaccination | Day 14 Post-Second Vaccination
  Measured using live-virus mpox neutralization assay, plaque reduction neutralization assay (PRNT).
Number of Solicited Adverse Events through Day 14 Post-Vaccinations | Day 14 Post-Vaccination
  Participants will complete a 14-day diary recording solicited adverse events following each vaccination.
Number of Adverse Events that Occur within 28 Days After Final Vaccination | Day 28 Post-Final Vaccination

SECONDARY OUTCOMES:
GMT of Mpox Virus-Specific Serum Immunoglobulin approximately 28 Days After First Vaccination | Day 28 Post-First Vaccination
  Measured using enzyme-linked immunosorbent assay (ELISA).
GMT of Mpox Virus-Specific Serum Immunoglobulin approximately 56 Days After First Vaccination | Day 56 Post-First Vaccination
  Measured using enzyme-linked immunosorbent assay (ELISA).
GMT of Mpox Virus-Specific Serum Immunoglobulin approximately 14 Days After Second Vaccination | Day 56 Post-Second Vaccination
  Measured using enzyme-linked immunosorbent assay (ELISA).
GMT of Serum Neutralization of Mpox Virus approximately 28 Days After First Vaccination | Day 28 Post-First Vaccination
  Measured using live-virus mpox neutralization assay, plaque reduction neutralization assay (PRNT).
GMT of Serum Neutralization of Mpox Virus approximately 56 Days After First Vaccination | Day 56 Post-First Vaccination
  Measured using live-virus mpox neutralization assay, plaque reduction neutralization assay (PRNT).

CONTACTS AND LOCATIONS:
Overall Officials: Angelica Kottkamp, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Dr. Mark Mulligan at 877-919-2822. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Dr. Mark Mulligan at 877-919-2822. To gain access, data requestors will need to sign a data access agreement.